CLINICAL TRIAL: NCT05131633
Title: Point-of-care Regional Anaesthesia in Intensive Care Unit. A Multicentric Professional Practice Evaluation
Brief Title: Regional Anaesthesia in Intensive Care Unit
Acronym: Week'ALR
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Hôpital Edouard Herriot (Other); Rangueil Hospital (Other); Hospices Civils de Lyon (Other); Hopital Louis Pradel (Other); Hôpital Saint Camille (Unknown); Hôpital de la Timone (Other); University Hospital, Grenoble (Other); University Hospital, Lille (Other); Saint Antoine University Hospital (Other); University Hospital, Strasbourg (Other); University Hospital, Marseille (Other); Centre Hospitalier Universitaire de Nīmes (Other); CH Aix (Unknown); CH Martigues (Unknown); CH Alberville (Unknown); CH Chambery (Unknown); Rennes University Hospital (Other); Bichat Hospital (Other)
Responsible Party: Principal Investigator, Blondonnet Raïko, Dr, University Hospital, Clermont-Ferrand
Other Study IDs: WEEK'ALR
Record Dates: First submitted 2021-10-03; First posted 2021-11-23 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Intensive Care Unit
Keywords: regional anesthesia; intensive care unit; analgesia; pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pain is a major problem in Intensive Care Unit (ICU). Adequate pain management not only means decreasing the pain intensity, but also improving the functionality and allowing the early mobilization that is a prerequisite for improving recovery and decreasing the risk of complications in ICU. The complex problems involved in pain, analgesic interventions, and outcome have been emphasized in several surveys over the past decades, but apparently with only small improvements, despite the existence of several guidelines for perioperative pain management.

Regional analgesia techniques (peripheral and neuraxial nerve blocks) have the potential to decrease the physiological stress response to trauma or surgery, reducing the possibility of surgical complications and improving the outcomes. Recent studies suggested that surgical and trauma ICU patients receive opioid-hypnotics continuous infusions to prevent pain and agitation that could increase the risk of posttraumatic stress disorder and chronic neuropathic pain symptoms, and chronic opioid use. Also they may reduce the total amount of opioid analgesics necessary to achieve adequate pain control and the development of potentially dangerous side effects. The use of the regional anesthesia technique in the ICU, however, can, in part, be limited by the presence of hemodynamic instability, bleeding diathesis, and by the fear of the performing procedures potentially associated with significant side effects in heavily sedated patients.

Although regional anesthesia emerges as a new and very interesting player for pain management in ICU, today very few data exists about the use of RA (including PNB and neuraxial nerves blocks) by the practicians in ICU/stepdown units. The main objective of this study is to assess the use of RA for pain management both initiates in the operative room for surgical patients then transferred in ICU/stepdown units and performs directly by the practicians in ICU/stepdown units, in several french units.

DETAILED DESCRIPTION:
Taken together, previous data indicate that regional anesthesia emerges as a new and very interesting player for pain management in ICU.

Because very few data exist about the use of RA (including PNB and neuraxial nerves blocks) by the practicians in ICU we, therefore, design this multicentric professional practice evaluation to :

* (1) , assess the use of RA in ICU/stepdown units but initiates by anesthesiologist in the operative room
* (2) , assess the use of RA in ICU/stepdown units directly perform by practicians in ICU
* (3) , describe the type, modalities and indications of RA performed

This study will have no effect on the management of the ICU/stepdown units patients.

ELIGIBILITY:
Inclusion Criteria:

○ All medical, surgical, and trauma patients hospitalized in the participating centers and receiving RA during the one-week study period.

Exclusion Criteria:

* Opposition to the processing of personal data
* Age <18 years old
* Absolute contraindications to the perform RA
* Previous hypersensitivity or anaphylactic reaction to local anesthetics
* Patient under a tutelage measure or placed under judicial protection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All medical, surgical, and trauma patients hospitalized in the participating centers and receiving RA during the one-week study period.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Our primary objective is to assess the global use of RA in ICU/stepdown units | During 1 week of the study
  . Number (prevalence) of RA performed in ICU over 1 week.

SECONDARY OUTCOMES:
assess the use, in ICU/stepdown units patients, of RA previously initiated in the operative room by an anesthesiologist | During 1 week of the study
  .Number of RA performed in operative room and then transferred in ICU over a week.
  . Prevalence of RA performed in the operative room and then transferred in ICU over a week
Type of RA | During 1 week of the study
  Nerves block or spinal anesthesia or epidural anesthesia
Location of RA | During 1 week of the study
  ICU or step-down unit or operating room
Who perform RA | During 1 week of the study
  Resident or senior and intensivist or anesthesiologist
Name of local anesthetics used | During 1 week of the study
  Name of local anesthetics used
Concentration of local anesthetics used | During 1 week of the study
  Concentration in mg/ml
Indications for RA | During 1 week of the study
  Analgesia or anesthesia or mobilization or nursing or weaning from mechanical ventilation
Technical management to perform RA | During 1 week of the study
  Type of needle
Technical management to perform RA | During 1 week of the study
  Use of sonography (yes / no)
Technical management to perform RA | During 1 week of the study
  Use of electrical nerve stimulator (yes / no)
Technical management to perform RA | During 1 week of the study
  Use of continuous catheter (yes / no)
Evaluation of analgesia | During 1 week of the study
  Visual Analog Score for pain)
Evaluation of success or not in RA | During 1 week of the study
  Sensitive and/or motor block
Contraindication for RA | During 1 week of the study
  Type of contraindication
Complication of RA | During 1 week of the study
  Type of complication
Reason for removal cathete | During 1 week of the study
  Type of reason
Duration of catheter | During 1 week of the study
  Duration in days
ICU/stepdown units length of stay | Day 28 after the RA
  Length in days
Hospital length of stay | Day 28 after the RA
  Length in days
Evaluation of vital status: on ICU/stepdown units discharge | Day 28 after the RA
Evaluation of vital status at day 28 | Day 28 after the RA
  Death or alive
Ventilator-free days to day 28 | Day 28 after the RA
  Unit : days

CONTACTS AND LOCATIONS:
Overall Officials: Raïko Blondonnet, Principal Investigator — rblondonnet@chu-clermontferrand.fr
Locations (19):
- France (19):
  - CH, Aix-en-Provence
  - CH, Bry-sur-Marne
  - CH, Chambéry
  - CHU, Clermont-Ferrand
  - Centre Jean-Perrin, Clermont-Ferrand
  - CHU, Grenoble
  - CHU, Lille
  - HCL Centre des Grands Brulés, Lyon
  - HCL Hôpital Sud, Lyon
  - APHM la Timone, Marseille
  - APHM Nord, Marseille
  - CHU, Nîmes
  - AHPH Saint-Antoine, Paris
  - APHP Bichat, Paris
  - CHU, Reims
  - CHU, Rennes
  - CH, Saint-Grégoire
  - CHU, Strasbourg
  - CHU, Toulouse